CLINICAL TRIAL: NCT03286829
Title: A Randomized, Open-label, Single-dose, Parallel-arm, Phase 1 Study to Investigate the Pharmacokinetic Profile of a Fixed-Dose Combination Tablet of Tesofensine and Metoprolol (Tesomet) and Co-Administration of Tesofensine Plus Commercial Metoprolol in Adult Healthy Subjects
Brief Title: Study to Investigate the Pharmacokinetic Profile
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TM003
Record Dates: First submitted 2017-09-05; First posted 2017-09-19 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tesomet "High dose" in fasted condition (Experimental): A Tesomet FDC tablet (20 mg immediate release [IR] metoprolol, 1 mg tesofensine, 80 mg extended release [ER] metoprolol) in fasted condition ("High" dose)
  Interventions: Drug: Comperator 1 mg tesofensine, 25 mg commercial IR metoprolol, 75 mg commercial ER metoprolol, fasted condition.
- Tesomet "Low dose" in fasted condition (Experimental): Treatment B (Test 2): A Tesomet FDC tablet (5 mg immediate IR metoprolol, 0.2 mg tesofensine, 20 mg ER metoprolol) in fasted condition. ("Low" dose)
  Interventions: Drug: Comperator 1 mg tesofensine, 25 mg commercial IR metoprolol, 75 mg commercial ER metoprolol, fasted condition.
- Comperator (Active Comparator): 1 mg tesofensine (2 tablets of 0.5 mg), 25 mg commercial IR metoprolol (1 tablet of 25 mg), 75 mg commercial ER metoprolol (1 tablet of 25 mg ER metoprolol and 1 tablet of 50 mg ER metoprolol), fasted condition
  Interventions: Drug: Tesomet "High dose" in fasted condition; Drug: Tesomet "Low dose" in fasted condition; Drug: Tesomet "High dose" in fed condition
- Tesomet "High dose" in fed condition (Experimental): A Tesomet FDC tablet (20 mg immediate IR metoprolol, 1 mg tesofensine, 80 mg ER metoprolol in fed condition ("High" dose)
  Interventions: Drug: Tesomet "High dose" in fasted condition; Drug: Comperator 1 mg tesofensine, 25 mg commercial IR metoprolol, 75 mg commercial ER metoprolol, fasted condition.

INTERVENTIONS:
Drug: Tesomet "High dose" in fasted condition — To evaluate the PK profile and relative bioavailability of a single dose of the Tesomet fixed-dose combination (FDC) tablet and co-administration of tesofensine plus commercial metoprolol.
  Other Names: Tesofensine; Metoprolol
  Arms: Comperator; Tesomet "High dose" in fed condition
Drug: Tesomet "Low dose" in fasted condition — To evaluate the PK profile and relative bioavailability of a single dose of the Tesomet fixed-dose combination (FDC) tablet and co-administration of tesofensine plus commercial metoprolol.
  Other Names: Tesofensine; Metoprolol
  Arms: Comperator
Drug: Comperator 1 mg tesofensine, 25 mg commercial IR metoprolol, 75 mg commercial ER metoprolol, fasted condition. — To evaluate the PK profile and relative bioavailability of a single dose of the Tesomet fixed-dose combination (FDC) tablet and co-administration of tesofensine plus commercial metoprolol.
  Other Names: Tesofensine; Metoprolol
  Arms: Tesomet "High dose" in fasted condition; Tesomet "High dose" in fed condition; Tesomet "Low dose" in fasted condition
Drug: Tesomet "High dose" in fed condition — To evaluate the PK profile and relative bioavailability of a single dose of the Tesomet fixed-dose combination (FDC) tablet and co-administration of tesofensine plus commercial metoprolol.
  Other Names: Tesofensine; Metoprolol
  Arms: Comperator

SUMMARY:
A randomized, open-label, single-dose, parallel-arm, Phase 1 study to investigate the pharmacokinetic profile of a fixed-dose combination tablet of tesofensine and metoprolol (Tesomet) and co-administration of tesofensine plus commercial metoprolol in adult healthy subjects

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel-arm study in 60 healthy male subjects who meet the inclusion and none of the exclusion criteria for the study. Each subject will participate in a screening period, a baseline period (the day preceding drug administration), and a single-dose treatment period with an on-site observation period of at least 48 hours after the dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the Screening Visit procedures.
2. Males between 18 to 55 years of age, inclusive, at the Screening Visit.
3. Nonsmokers (or other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (< 500 ng/mL) at the Screening Visit and admission.
4. BMI between 18.5 and 30.0 kg/m2, inclusive, at the Screening Visit.
5. Healthy, determined by pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory evaluations).

Exclusion Criteria:

1. Subject has history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy as judged by the Investigator.
2. Subject has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Subject has history of alcohol and/or illicit drug abuse within 2 years of entry.
4. Subject is unwilling to avoid consumption of coffee and caffeine-containing beverages within 48 hours prior to admission until discharge from the clinical site.
5. Subject is unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to admission until discharge from the clinical site.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen Drejer, PhD, Study Director — Saniona
Locations (1):
- Early Phase Clinical Unit;Klinikum Westend, Haus 31, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tesomet "Low Dose" in Fasted Condition: A Tesomet FDC tablet (5 mg immediate IR metoprolol, 0.2 mg tesofensine, 20 mg ER metoprolol) in fasted condition. ("Low" dose)
- Comparator: 1 mg tesofensine (2 tablets of 0.5 mg), 25 mg commercial IR metoprolol (1 tablet of 25 mg), 75 mg commercial ER metoprolol (1 tablet of 25 mg ER metoprolol and 1 tablet of 50 mg ER metoprolol), fasted condition
Period: Overall Study
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tesomet "High Dose" in Fasted Condition: Tesomet FDC tablet (20 mg immediate release [IR] metoprolol, 1 mg tesofensine, 80 mg extended release [ER] metoprolol) in fasted condition ("High" dose)
- Tesomet "Low Dose" in Fasted Condition: Tesomet FDC tablet (5 mg immediate IR metoprolol, 0.2 mg tesofensine, 20 mg ER metoprolol) in fasted condition. ("Low" dose)
- Tesomet "High Dose" in Fed Condition: Tesomet FDC tablet (20 mg immediate IR metoprolol, 1 mg tesofensine, 80 mg ER metoprolol in fed condition ("High" dose)
- Total: Total of all reporting groups
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 40.3 (11.55) | 41.1 (8.81) | 39.5 (10.19) | 41.9 (9.91) | 40.7 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 15 | 15 | 15 | 15 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 15 | 15 | 59
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 14 | 15 | 15 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: AUC0-48
Description: Area under the concentration-time curve from pre-dose (time 0) to 48 hours post-dose calculated using the linear-log trapezoidal rule
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30, 36 and 48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng*hr/mL | 32.06 (26.9) | 6.491 (25.1) | 45.89 (21.9) | 30.14 (18.6)

2. Secondary Outcome: Cmax
Description: Maximum tesofensine and metoprolol concentrations determined directly from the concentration-time profile
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30, 36 and 48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/mL | 0.9528 (25.5) | 0.1934 (23.6) | 1.357 (23.8) | 0.8085 (17.1)

3. Secondary Outcome: Tmax
Description: Time of maximum tesofensine and metoprolol concentrations determined directly from the concentration-time profile
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 30, 36 and 48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition
Number analyzed (Participants) | 15 | 15 | 15 | 15
hours | 6.12 (5.98) | 6.00 (5.98) | 6.00 (3.98) | 8.00 (4.00)

ADVERSE EVENTS:
Time Frame: 38days
Arm/Group | Tesomet "High Dose" in Fasted Condition | Tesomet "Low Dose" in Fasted Condition | Comparator | Tesomet "High Dose" in Fed Condition
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 4/15 | 5/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3.33% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesomet "High Dose" in Fasted Condition (N=15) | Tesomet "Low Dose" in Fasted Condition (N=15) | Comparator (N=15) | Tesomet "High Dose" in Fed Condition (N=15)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
catheter side reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03286829/Prot_000.pdf
  • Informed Consent Form (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03286829/ICF_001.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT03286829/SAP_002.pdf